CLINICAL TRIAL: NCT03955627
Title: Using Exercise to Relieve Arthralgia (Joint Pain) and Improve AI Adherence in Older Survivors (REJOIN): A Pilot Study
Brief Title: REJOIN Trial for Older Breast Cancer Survivors
Acronym: REJOIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00089191; 40010042 (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2019-04-29; First posted 2019-05-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Female
Keywords: Cancer Treatment Symptoms, Symptom Management

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Pilot. Enhanced Standard Care v. Treatment (education plus exercise).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Masked parties will not be told the arm to which the participant is assigned. Patient study records will indicate if they are in the study, but not the arm assignment. All participants will receive standard information about AI use and participate in four assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Standard Care (No Intervention): Participants will receive standard care, plus a brochure about hormonal therapy use.
- Treatment (Education plus Exercise) (Experimental): Participants will receive the same materials as the standard care group, plus participate in group exercise and group discussion sessions.
  Interventions: Behavioral: Relieving Joint Pain and Improving AI Adherence in Older Breast Cancer Survivors (REJOIN)

INTERVENTIONS:
Behavioral: Relieving Joint Pain and Improving AI Adherence in Older Breast Cancer Survivors (REJOIN) — Self-management program which includes supervised exercise sessions in groups and group discussions for 8 weeks conducted by Zoom video, followed by an 8-week home-based version of the same program participants do on their own with bi-weekly coaching calls.
  Other Names: REJOIN
  Arms: Treatment (Education plus Exercise)

SUMMARY:
The purpose of this pilot intervention study is to test the effectiveness of a self-management approach (combining education- and exercise-based strategies) for improving arthralgia (joint pain) associated with Aromatase Inhibitors (AI) in older breast cancer survivors. Survivors will be recruited from local cancer clinics prior to the completion of primary cancer treatment, as arthralgia can occur soon after initiating AI medication. Participants will be randomized to one of two groups: an enhanced standard care group (AI prescription plus information) or a treatment group (educational classes plus group exercise sessions). Older survivors (≥60 years) will be targeted because they are at increased risk of medication complications which may impede adherence. For the baseline assessment, a cancer-specific geriatric assessment will be conducted and a blood sample will be collected to interpret the effects of the self-management study in the context of geriatric experiences. Additionally, there will be an assessment of knowledge, PA habits, and AI-related joint pain and AI adherence. These will be measured again at 4, 6 and at follow up at 12 months.

DETAILED DESCRIPTION:
To improve AIA and AI Adherence in older survivors, it will: first, adapt an evidence-based intervention (AIM 1) and then; test the adapted intervention with breast cancer survivors ≥65 years. The Investigators will educate survivors about possible AI-related side effects and teach survivors ways to use PA to self-manage AIA (AIM 2), and support adherence to hormonal therapy recommendations (AIM 3). Given evidence that survivors experience AIA soon after initiating hormonal therapy, potentially eligible participants would be identified early in the treatment process. By identifying potential participants after diagnosis or during active treatment, survivors would have a minimal delay in beginning the exercise intervention after initiating hormonal therapy (i.e. AIs). All participants will have completed surgery, radiation and/or chemotherapy, which is consistent with current ASCO guidelines for AI use.

Two groups will be randomized to either an information-only group (enhanced standard care) or an education plus exercise group (treatment). At the initial clinical visit during the intervention, participants in both groups will receive printed information along with their AI medication prescription. The treatment group will subsequently receive a one-on-one exercise consultation with a certified exercise trainer (e.g ACSM or similar), followed by a modified version of the Fit & Strong! program, which includes bi-weekly supervised exercise (60 minutes) and educational sessions (30 minutes).

The exercise sessions will include light weights or resistance bands plus low-impact aerobic exercise, in which movements will be explained, demonstrated and modified based on the needs of participants. The exercise protocol will be reviewed and revised based on recommendations from clinical advisers. Educational materials will provide information about the purpose of AI medications (e.g., to reduce cancer recurrence) in layperson language and basic information about potential side effects. As part of in-person sessions, participants will develop a plan to continue exercise at home. Participants can do an activity of their choice (e.g., walking) and use resistance bands which will be provided for the at-home program which will begin after 8 weeks and will include follow up phone calls to assess progress and reinforce the program. Educational sessions will be modified to reflect relevant content and advice for older survivors beginning AIs. Assessments will be taken at 4 and 6 months, with follow up at 12 months.

All supervised exercise sessions will be conducted remotely to accommodate recommended COVID safety protocols.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged ≥ 60 years at the start of study
* Planning to initiate AIs
* Diagnosed stages I-III Breast Cancer
* R+ tumor (at least 5% of cells)
* Completed surgery, radiation and/or chemotherapy
* Independent ambulatory (verified by treating clinician/staff)
* Physician approval to start an exercise program
* Must report insufficient physical activity (<150 min. of physical activity per week)
* Able to complete surveys and forms/ understand English
* Agree to random assignment to exercise or control group
* Can commit to 8 weeks, bi-weekly classes offered by Zoom video
* Must have internet access and/or data plan by which to participate in Zoom video sessions
* Minimum cognitive impairment (verified by cognitive screening questions administered by phone or in-person interview)

Exclusion Criteria:

* Already taking Aromatase Inhibitors (AIs) (may participate if 24 weeks or less after initiating)
* Presence of metastatic cancer or concurrent malignancy requiring treatment
* Recent history (past 6 months) of stroke/ Myocardial Infarction (MI), atrial fibrillation or class 3, 4 heart failure
* Recent joint surgery or conditions limiting PA

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be biologically female
Enrollment: 12 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Change in Brief Pain Inventory (Modified for Joint Pain) Scores | baseline at 12 months
  The Brief Pain Inventory - Short Form (BPI-sf) is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale. The BPI-sf is a modification of the Brief Pain Inventory - Long Form, which includes additional questions on demographics (date of birth, marital status, education, employment), pain history, aggravating and easing factors, treatment and medication, pain quality, and response to treatment. Higher scores indicate greater severity and more interference.

SECONDARY OUTCOMES:
AI Medication Adherence Percentage | Day 30
  Medication Possession Ratio (MPR). Percent of days medication taken as prescribed, as self-reported by patient and verified with prescription refill records.
Change in Toronto Informational Needs Questionnaire (TINQ) Scores -- Breast Cancer | Month 12
  Self-report questionnaire about knowledge of breast cancer, its treatment and its side effects. Responses to questions about informational needs are reported using a Likert Scale -- 1 is "not important" to 5 "extremely important." Higher score indicate greater informational needs. Individual subscales may be calculated using percentages.
Change in Modified Cancer and Aging Research Group (CARG) plus National Health and Nutrition Examination Survey (NHANES) and Patient-Reported Outcomes Measurement Information System (PROMIS) Geriatric Assessment Study Patient Questionnaire | Month 12
  Aggregated assessment of self-reported information about demographic data, daily activities, nutritional status, medication use and health behaviors.
Change in Community Healthy Activities Model Program for Seniors (CHAMPS) Questionnaire Scores for Older Adults | Month 12
  This self-report questionnaire assesses weekly frequency and duration of a variety of lifestyle physical activities that are meaningful and appropriate for older adults. It includes activities of various intensities (from light to vigorous) such as walking, running, hiking, swimming, bicycling, dancing, tennis, aerobics, yoga/tai chi, gardening, and housework. Intensity is reflected in the item stem (e.g., light and heavy gardening are separate items).
Change in Exercise Self-efficacy Scale Scores | Month 12
  The Exercise Self-Efficacy Scale assesses an individual's beliefs in their ability to continue exercising on a three time per week basis at moderate intensities for 40+ minutes per session in the future. For each of 8 items, participants indicate their confidence to execute the behavior on a 100-point percentage scale comprised of 10-point increments, ranging from 0% (not at all confident) to 100% (highly confident). Total strength for each measure of self-efficacy is then calculated by summing the confidence ratings and dividing by the total number of items in the scale, resulting in a maximum possible efficacy score of 100.
Inflammatory biomarker amounts | Baseline and Month 12
  Fasting blood sample (2 tsp) to assess inflammatory biomarkers (IL-6, TNFα, C-reactive protein [CRP])

CONTACTS AND LOCATIONS:
Overall Officials: Shirley M Bluethmann, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We will share deidentified data only, if requested.

REFERENCES:
- [Derived] Bluethmann SM, Truica C, Klepin HD, Olsen N, Sciamanna C, Chinchilli VM, Schmitz KH. Study design and methods for the using exercise to relieve joint pain and improve AI adherence in older breast cancer survivors (REJOIN) trial. J Geriatr Oncol. 2021 Sep;12(7):1146-1153. doi: 10.1016/j.jgo.2021.05.011. Epub 2021 May 26. PMID 34049837

DOCUMENTS (1):
  • Informed Consent Form (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT03955627/ICF_000.pdf